CLINICAL TRIAL: NCT04402411
Title: Comparison Between Quadratus Lumborum Block and Transversus Abdominis Plane Block in Bladder Cancer Surgeries
Brief Title: Quadratus Lumborum Block vs Transversus Abdominis Plane Block in Bladder Cancer Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201617049.3
Record Dates: First submitted 2020-04-18; First posted 2020-05-26 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Quadratus Lumborum Block; Transversus Abdominis Plane Block; Bladder Cancer; Postoperative Pain; Surgery
MeSH Terms: conditions — Urinary Bladder Neoplasms; Pain, Postoperative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): Patients will receive general anesthesia with intravenous opioid
  Interventions: Drug: Intravenous opioid
- Quadratus lumborum (Experimental): Patients will receive bilateral quadratus lumborum block
  Interventions: Procedure: Quadratus lumborum block
- Transversus abdominis plane (Experimental): Patients will receive bilateral transversus abdominis plane block
  Interventions: Procedure: Transversus abdominis plane block

INTERVENTIONS:
Procedure: Quadratus lumborum block — The patient will be placed in a lateral position with the side to be blocked facing upwards. The ultrasound probe will be properly sterilized and with sterile covers. An 18-20 gauge blunt tipped block needle or a Tuohy needle is advanced under ultrasound guidance on the posterior aspect of the Quadratus Lumborum. The QL muscle is identified with its attachment to the lateral edge of the transverse process of the L4 vertebral body. With the psoas major muscle anteriorly, the erector spinae muscle posteriorly and the QL muscle adherent to the apex of the transverse process, a well recognisable pattern of a shamrock with three leaves can be seen.
  Other Names: Group B
  Arms: Quadratus lumborum
Procedure: Transversus abdominis plane block — The patient will be supine while performing the block and sterilization of the site of the ultrasound and needle entry will be performed.
  The ultrasound probe is placed in a transverse plane to the lateral abdominal wall in the midaxillary line, between the lower costal margin and iliac crest.
  The needle is introduced in plane of the ultrasound probe directly under the probe and advanced until it reaches the plane between the internal oblique and transversus abdominis muscles.
  Other Names: Group C
  Arms: Transversus abdominis plane
Drug: Intravenous opioid — Patients will receive morphine 0.1 mg/kg
  Other Names: Group A
  Arms: Control Group

SUMMARY:
Transversus abdominis plane (TAP) block can be used to provide effective analgesia during the postoperative period following a range of surgeries.

TAP block administers local anesthetics between the T6 to L1 spinal nerve roots to stop the nerve signal and to alleviate pain for abdominal procedures 4, 5.

The viscera are innervated by the vagal nerve (parasympathetic innervation) and by the splanchnic nerves (sympathetic innervation). The splanchnic nerves carry both visceral efferent and afferent nerve fibers. The sensory (or afferent) part of the splanchnic nerves reach the spinal column at certain spinal segments, It is possible to block central visceral pain conduction with thoracic paravertebral blockade or maybe even with the novel quadratus lumborum (QL) block.

The effect of the QL block is believed to result from a spread of LA from its lumbar deposition cranially into the thoracic paravertebral space (TPVS), since Carney et al found traces of contrast agent in the TPVS following application of this block. Hence, the QL block would seem to be able to alleviate both somatic and visceral pain.10

The aim of this study is to compare between quadratus lumborum block, transversus abdominis plane block regarding perioperative analgesia after bladder cancer surgeries by measuring intraoperative hemodynamics, postoperative pain scores and morphine consumption in the first 24 h postoperative.

DETAILED DESCRIPTION:
Somatic post-surgical pain is very distressing to patients which leads to important complications. Combined multimodal strategies involving nerve blocks, neuroaxial blocks, opiates, and non-steroidal anti-inflammatory drugs are necessary for optimal pain control.

Transversus abdominis plane (TAP) block can be used to provide effective analgesia during the postoperative period following a range of surgeries.

TAP block administers local anesthetics between the T6 to L1 spinal nerve roots to stop the nerve signal and to alleviate pain for abdominal procedures.

A number of systematic reviews have assessed TAP block as a postoperative analgesic compared to one or more specific procedures.

Anterior abdominal wall blocks, as transverse abdominal plexus block, have an important role for only somatic intraoperative and postoperative pain control.

The viscera are innervated by the vagal nerve (parasympathetic innervation) and by the splanchnic nerves (sympathetic innervation). The splanchnic nerves carry both visceral efferent and afferent nerve fibers. The sensory (or afferent) part of the splanchnic nerves reach the spinal column at certain spinal segments, It is possible to block central visceral pain conduction with thoracic paravertebral blockade or maybe even with the novel quadratus lumborum (QL) block.

The effect of the QL block is believed to result from a spread of LA from its lumbar deposition cranially into the thoracic paravertebral space (TPVS), since Carney et al found traces of contrast agent in the TPVS following application of this block. Hence, the QL block would seem to be able to alleviate both somatic and visceral pain.10 Quadratus lumborum block was first described by Blanco in 2007. Blanco described a potential space posterior to the abdominal wall muscles and lateral to the quadratus lumborum muscle. It has been used in abdominoplasties, caesarean sections and lower abdominal operations providing complete pain relief in the distribution area from Th6 to L1 dermatomes. It may be seen as a lumbar approach to the Thoracic Paravertebral Space. The block apparently produces distribution of the local anesthetic extending proximally and over both sides of the surface of the QL muscle, in between the anterior and intermediate layers of the thoracolumbar fascia.

Quadratus lumborum muscle inserts on the lower border of the last rib and by four small tendons into the apices of the transverse processes of the upper four lumbar vertebrae.

Running between its fascia and the muscle are the twelfth thoracic (subcostal), ilioinguinal, and iliohypogastric nerves, The block does not rely on the feeling of any pops or fascial clicks because depending of the angle of the needle several pops can be felt without reaching the target zone, which is lateral to the quadratus lumborum muscle. Actually, the block has never been intended to be conducted without the use of US guidance, and the block is thus a purely USG block.

Aim of study Comparison between quadratus lumborum block, transversus abdominis plane block regarding perioperative analgesia after bladder cancer surgeries by measuring intraoperative hemodynamics, postoperative pain scores and morphine consumption in the first 24 h postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Age of the patients between 20 to 80 years.
* ASA physical status II -III
* Elective bladder cancer operations.

Exclusion Criteria:

* Patient refusal
* Local infection at the site of injection
* Allergy to study medications
* Sepsis
* Anatomic abnormalities
* Systemic anticoagulation or coagulopathy
* Inability to comprehend or participate in pain scoring system

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-05 (Estimated)

PRIMARY OUTCOMES:
Time to first rescue dose of morphine | 24 hours
  First time at which morphine was given postoperatively (If Vsual analogue scale (VAS) was >4, 3 mg morphine IV was administered as a rescue analgesia for the first 24 hours)

SECONDARY OUTCOMES:
Total dose of postoperative morphine consumption | 24 hours
  Postoperative analgesia was provided by 1 gm paracetamol IV every 8 hours as a routine analgesia and if VAS was >4, 3 mg morphine IV was administered as a rescue analgesia for the first 24 hours.
Pain intensity by visual analogue scale (VAS) | 24 hours
  Visual analogue scale (VAS) was recorded at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24 hours postoperative.
  (0: No pain, 1-3: Mild pain, 4-6: Moderate pain, 7-9: Severe pain and 10: The worst imaginable pain) Minimum:0 and Maximum 10 The higher, the worst

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Mohammed, MSc, Principal Investigator — Assistant lecturer of Anesthesia, ICU, and Pain Relief
Locations (1):
- National Cancer Institute - Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
I don't want to share